CLINICAL TRIAL: NCT06700967
Title: A Precision Medication Guidance Model for Schizophrenia Based on Pharmacogenomics and Physiologically Based Pharmacokinetics: a Real-World Observational Study
Brief Title: Evaluating Pharmacogenomics-Based Pharmacotherapy in Real-World Settings for Schizophrenia
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: CRC2021ZD02
Record Dates: First submitted 2024-10-23; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Schizophenia Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An 8-week, rater-blinded, real-world observational study to investigate the benefits of pharmacogenetics-based pharmacotherapy in patients suffering from schizophrenia.

DETAILED DESCRIPTION:
This study, conducted at the Shanghai Mental Health Center, aims to compare changes in treatment efficacy and the frequency and severity of adverse reactions in patients with schizophrenia who have experienced treatment failure, before and after implementing a pharmacogenomics-based precision medication guidance strategy. The research is set in real-world conditions, without a predetermined treatment regimen for participants; instead, medication optimization is guided by pharmacogenomic testing results. Following the receipt of precision medication recommendations for each participant, the study physicians optimize the treatment regimen based on these recommendations and their clinical expertise. Optimization may involve adjusting the dose of current medications (if the existing regimen is largely suitable), switching medications (in cases of inappropriate treatment), or modifying the dose or replacing one of the combined medications (to manage drug-drug interactions). The rationality of the medication regimen will be assessed at the end of weeks 4 and 8, with additional recommendations provided as needed. Treatment effectiveness and safety will be evaluated during follow-up visits at these intervals. A total of 400 patients are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Suffer from schizophrenia (as assessed in agreement with ICD-11 criteria).
2. Age between ≥18 and <65 years.
3. Currently receiving inpatient or outpatient psychiatric treatment.
4. Experienced any of the following suboptimal treatment conditions while receiving antipsychotic medication within the therapeutic dosage range:

   1. Standard antipsychotic treatment for more than 2 weeks with the occurrence of drug-induced adverse effects requiring dose adjustment or a switch of medication.
   2. Antipsychotic treatment within the therapeutic dosage range for more than 4 weeks, with the presence of at least two items of the Positive and Negative Syndrome Scale (PANSS) (P1, P2, P3, N1, N4, N6, G5, and G9) score ≥4, or a total PANSS score >70, or a CGI-S score ≥4.
   3. Other situations where a change in medication is deemed necessary, as assessed by senior clinical physicians.
5. Understand the study requirements and provide written informed consent to participate; a signed and dated informed consent form (ICF) will be obtained from each patient before participation in the study.

Exclusion Criteria:

1. Presence of organic brain disease or a severe and/or unstable physical condition.
2. Substance abuse or dependence within the past 6 months or currently.
3. Presence of elevated levels of agitation, impulsivity, or risk of self-injury or suicide.
4. Pregnant or breastfeeding women.
5. The presence of any other conditions that may render the individual ineligible for participation in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes outpatients or inpatients receiving treatment at the Shanghai Mental Health Center in Shanghai, China
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Total Score at Week 4 and Week 8 | 4 weeks and 8 weeks
  The Positive and Negative Syndrome Scale (PANSS) provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme). It's designed to capture symptoms of schizophrenia. Score range 30-210. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Change in the Calgary Depression Scale for Schizophrenia (CDSS) | 4 weeks and 8 weeks
  The Calgary Depression Scale for Schizophenia (CDSS) is a 9-item scale used to rate the depressive symptoms in patients with schizophrenia. For each CDSS item, symptom severity was rated on a 3-point scale, from 0=absent to 3=severe. The CDSS total score ranges from 0 to 27 with a higher score indicating a greater severity of symptoms.
Change in the Clinical Global Impression of Severity (CGI-S) | 4 weeks and 8 weeks
  The Clinical Global Impression of Severity (CGI-S) rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale. It is rated as follows: 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Among the most extremely ill. Higher scores indicate worsening
Clinical Laboratory Tests | 4 weeks and 8 weeks
  Test data of the Hematology, Serum chemistry, Lipid Panel, Glycated Hemoglobin, Urinalysis, etc. will be collocted.
Safety Assessment by the Treatment Emergent Symptom Scale (TESS) score | 4 weeks and 8 weeks
  The Treatment Emergent Symptom Scale (TESS) consists of behavioral toxicity, laboratory abnormalities, nervous system, automatic nervous system, cardiovascular system and six other aspects, was used to evaluate adverse drug reactions based on the scores, ranging from 0 to 4 (the higher the score, the more serious the adverse reactions).
Safety Assessment by Barnes Akathisia Rating Scale(BARS) | 4 weeks and 8 weeks
  BARS consisted of 4 items, and the first 3 items were rated on a 4-point scale: 0 = absence of symptoms to 3 = severe condition. The global clinical evaluation was made on a 6-point scale, (0=absent, 1=questionable, 2=mild, 3=moderate, 4=marked, 5=severe). The BARS Global Score was derived from the global clinical assessment of akathisia from the BARS panel. The total score ranges from 0 to 14. The higher number indicates a worse outcome.
Safety Assessment by Simpson-Angus Scale(SAS) | 4 weeks and 8 weeks
  The minimum of each item (Gait, Arm Dropping, Shoulder Shaking, Elbow Rigidity, Fixation of Position or Wrist Rigidity, Leg Pendulousness, Head Dropping, Glabella Tap, Tremor, Salivation) in the SAS (Simpson-Angus Scale) is 0, and the maximum is 4. The minimum total score in the SAS is 0, and the maximum is 40. The higher number is worse outcome.
Safety Assessment by Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score | 4 weeks and 8 weeks
  The Abnormal Involuntary Movement Scale (AIMS) Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.

OTHER OUTCOMES:
Change in the Medication Satisfaction Questionnaire (MSQ) score | 8 weeks
  The medication satisfaction questionnaire (MSQ) is a single-item, global, patient-completed instrument that is read aloud to patients by clinicians designed to assess treatment satisfaction among patients with schizophrenia. It consists of one question: "Overall, how satisfied are you with your current antipsychotic medication(s)?" with responses assessed on a 7-point scale rated as follows: 1 = extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=neither satisfied nor dissatisfied, 5=somewhat satisfied, 6 = very satisfied, 7 = extremely satisfied.
Change in the Drug Attitude Inventory (DAI)-10 Score | 8 weeks
  DAI, a 10-item scale to assess how the attitude of schizophrenia patients toward their medications may affect compliance. Respondents indicate 'true' or 'false' for each item. An overall calculated score ranges from -10 to 10, where a positive score indicated a positive subjective response (compliant), whilst a negative score indicated non-compliance.
Change in the Personal and Social Performance Scale (PSP) | 8 weeks
  The PSP is a 100-point validated clinician-rated scale that assesses the degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviors rated on a 6-point scale (1=absent to 6=very severe). Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty), with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caudle KE, Sangkuhl K, Whirl-Carrillo M, Swen JJ, Haidar CE, Klein TE, Gammal RS, Relling MV, Scott SA, Hertz DL, Guchelaar HJ, Gaedigk A. Standardizing CYP2D6 Genotype to Phenotype Translation: Consensus Recommendations from the Clinical Pharmacogenetics Implementation Consortium and Dutch Pharmacogenetics Working Group. Clin Transl Sci. 2020 Jan;13(1):116-124. doi: 10.1111/cts.12692. Epub 2019 Oct 24. PMID 31647186
- [Background] Gaedigk A, Simon SD, Pearce RE, Bradford LD, Kennedy MJ, Leeder JS. The CYP2D6 activity score: translating genotype information into a qualitative measure of phenotype. Clin Pharmacol Ther. 2008 Feb;83(2):234-42. doi: 10.1038/sj.clpt.6100406. Epub 2007 Oct 31. PMID 17971818
- [Background] Kane JM, Kinon BJ, Forray C, Such P, Mittoux A, Lemming OM, Hertel P, Howes OD; DayBreak and Debut study investigators. Efficacy and safety of Lu AF35700 in treatment-resistant schizophrenia: A randomized, active-controlled trial with open-label extension. Schizophr Res. 2022 Oct;248:271-278. doi: 10.1016/j.schres.2022.09.012. Epub 2022 Sep 14. PMID 36115192
- [Background] Lindenmayer JP, Citrome L, Khan A, Kaushik S, Kaushik S. A randomized, double-blind, parallel-group, fixed-dose, clinical trial of quetiapine at 600 versus 1200 mg/d for patients with treatment-resistant schizophrenia or schizoaffective disorder. J Clin Psychopharmacol. 2011 Apr;31(2):160-8. doi: 10.1097/JCP.0b013e31820f4fe0. PMID 21346616
- [Background] Wojtyniak JG, Selzer D, Schwab M, Lehr T. Physiologically Based Precision Dosing Approach for Drug-Drug-Gene Interactions: A Simvastatin Network Analysis. Clin Pharmacol Ther. 2021 Jan;109(1):201-211. doi: 10.1002/cpt.2111. Epub 2020 Dec 6. PMID 33280091
- [Background] Hahn M, Roll SC. The Influence of Pharmacogenetics on the Clinical Relevance of Pharmacokinetic Drug-Drug Interactions: Drug-Gene, Drug-Gene-Gene and Drug-Drug-Gene Interactions. Pharmaceuticals (Basel). 2021 May 20;14(5):487. doi: 10.3390/ph14050487. PMID 34065361
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203